CLINICAL TRIAL: NCT05581355
Title: The Effect of Abdominal Breathing on Improving of Sleep Quality and Physiological Index Among Patients With Insomnia
Brief Title: Abdominal Breathing on Improving of Sleep Quality and Physiological Index Among Patients With Insomnia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Principal Investigator, Xuan-Yi Huang, RN, DNSc, Professor, National Taipei University of Nursing and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: (849)109A-88
Record Dates: First submitted 2022-09-28; First posted 2022-10-14 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Insomnia
Keywords: abdominal breathing; quality of sleep; physiological index; effectiveness
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: This study method adopts the research design of experimental randomized controlled trials. The persons receiving the intervention of abdominal breathing training are in the experimental group, while those who do not receive it are in the control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The effectiveness of receiving abdominal breathing training (Experimental): Training for 8 weeks (1 time a week, 15 minutes each time). Performed one-on-one by a trainer in a sleep center. At home, you can use the abdominal breathing training video to train yourself (10 minutes a day, can be divided into 10 minutes), and you need to fill in the abdominal breathing training log.
  Interventions: Behavioral: Abdominal breathing training
- The effectiveness of not receiving abdominal breathing training (No Intervention): The trainer does not provide abdominal breathing training, does not perform abdominal breathing exercises at home, and does not need to fill in abdominal breathing training logs.

INTERVENTIONS:
Behavioral: Abdominal breathing training — In the sleep center, it is carried out in a one-on-one manner by the trainer. At home, self-training through abdominal breathing training videos (10 minutes per day, you can accumulate up to 10 minutes in divided doses)
  Arms: The effectiveness of receiving abdominal breathing training

SUMMARY:
The research topic is to explore the effectiveness of abdominal breathing on improving of sleep quality and physiological index (heart rate, respiration rate and blood pressure) among patients with insomnia. This study method adopts the research design of experimental randomized controlled trials. The persons receiving the intervention of abdominal breathing training are in the experimental group, while those who do not receive it are in the control group.

DETAILED DESCRIPTION:
Sleep problem is very common symptom problems, so often rely on sedative-hypnotics drugs. However, long-term dependence on drugs may bring serious side effects. Therefore, the research topic is to explore the effectiveness of abdominal breathing on improving of sleep quality and physiological index (heart rate, respiration rate and blood pressure) among patients with insomnia. This study method adopts the research design of experimental randomized controlled trials. The persons receiving the intervention of abdominal breathing training are in the experimental group, while those who do not receive it are in the control group. The research is conducted with A and B groups. Group A is for those who take sedative and sleeping medicine, and Group B is for those who do not take sedative and sleeping medicine. Both groups A and B have experimental group and control group. The effectiveness assessment will use the Pittsburgh Quality Sleep Index (PSQI) and vital signs (heart rate, breathing and blood pressure). These assessments need to complete by both the experimental group and control group. This study uses the pre-test before the implementation of abdominal breathing training, and uses the post-test at week 4 and week 8 the end of abdominal breathing training. The experimental group will receive the abdominal breathing training for a total of 8 weeks. Abdominal breathing training is carry out in the sleep center of hospital (once every 1 week, and 15 minutes every time). When the persons are at home, they will receive self-training using the abdominal breathing training video (every day 10 minutes, can include every time during the day). Moreover, the persons need to complete the "abdominal breathing training log". Hopefully, this study may develop that does not use drugs, but improves sleep quality and physiological index through abdominal breathing.

ELIGIBILITY:
Inclusion Criteria:

* Those with a total score greater than 5 points on the Pittsburgh Sleep Product Quality Table have been diagnosed with insomnia based on the Taiwan Psychiatric Association (2014) DSM-5 Psychiatric Disorder Diagnosis and Statistics, who have agreed to participate in this study and have completed a written consent form.

Exclusion Criteria:

* Patients with COPD

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 138 (Actual)
Dates: Start 2021-01-14 (Actual); Primary Completion 2021-09-13 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index | Pre-test
  The total items of Pittsburgh Sleep Quality Index inventory are 7. The score of each item is from 0-3. The score>5 points means the sleep quality is good. Meanwhile the score ≦5 points is poor sleep quality.
Pittsburgh Sleep Quality Index | Post-test at week 4
  The total items of Pittsburgh Sleep Quality Index inventory are 7. The score of each item is from 0-3. The score>5 points means the sleep quality is good. Meanwhile the score ≦5 points is poor sleep quality.
Pittsburgh Sleep Quality Index | Post-test at week 8
  The total items of Pittsburgh Sleep Quality Index inventory are 7. The score of each item is from 0-3. The score>5 points means the sleep quality is good. Meanwhile the score ≦5 points is poor sleep quality.

SECONDARY OUTCOMES:
Heart rate | Pre-test
  Before the abdominal breathing record the heart rate
Respiration rate | Pre-test
  Before the abdominal breathing record the respiration rate
Blood pressure | Pre-test
  Before the abdominal breathing,record the blood pressure
Heart rate | Post-test at week 4
  After abdominal breathing for 4 weeks, and than record the heart rate
Respiration rate | Post-test at week 4
  After abdominal breathing for 4 weeks, and than record the respiration rate
Blood pressure | Post-test at week 4
  After abdominal breathing for 4 weeks, and than record the blood pressure
Heart rate | Post-test at week 8
  After abdominal breathing for 8 weeks, and than record the heart rate
Respiration rate | Post-test at week 8
  After abdominal breathing for 8 weeks, and than record the respiration rate
Blood pressure | Post-test at week 8
  After abdominal breathing for 8 weeks, and than record the blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Xuan-Yi Huang, DNSc, Principal Investigator — National Taipei University of Nursing and Health Sciences
Locations (1):
- Xuan-Yi Huang, Taipei, Peitou, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abad VC, Guilleminault C. Insomnia in Elderly Patients: Recommendations for Pharmacological Management. Drugs Aging. 2018 Sep;35(9):791-817. doi: 10.1007/s40266-018-0569-8. PMID 30058034
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Canham SL, Rubinstein RL. Experiences of sleep and benzodiazepine use among older women. J Women Aging. 2015;27(2):123-39. doi: 10.1080/08952841.2014.928173. Epub 2015 Jan 12. PMID 25581296
- [Background] Chen YF, Huang XY, Chien CH, Cheng JF. The Effectiveness of Diaphragmatic Breathing Relaxation Training for Reducing Anxiety. Perspect Psychiatr Care. 2017 Oct;53(4):329-336. doi: 10.1111/ppc.12184. Epub 2016 Aug 23. PMID 27553981
- [Background] Chennaoui M, Arnal PJ, Sauvet F, Leger D. Sleep and exercise: a reciprocal issue? Sleep Med Rev. 2015 Apr;20:59-72. doi: 10.1016/j.smrv.2014.06.008. Epub 2014 Jun 30. PMID 25127157
- [Background] de Jong AE, Gamel C. Use of a simple relaxation technique in burn care: literature review. J Adv Nurs. 2006 Jun;54(6):710-21. doi: 10.1111/j.1365-2648.2006.03858.x. PMID 16796663
- [Background] Hausler N, Marques-Vidal P, Haba-Rubio J, Heinzer R. Does sleep predict next-day napping or does napping influence same-day nocturnal sleep? Results of a population-based ecological momentary assessment study. Sleep Med. 2019 Sep;61:31-36. doi: 10.1016/j.sleep.2019.04.014. Epub 2019 May 4. PMID 31300205